CLINICAL TRIAL: NCT06229405
Title: Development of Clinical Evidence for Optimal Management of Adrenal Diseases Based on Real-World Data: An Initiative by the Korean Adrenal Disorder Study (KADS) Group
Brief Title: Development of Clinical Evidence for Optimal Management of Adrenal Diseases Based on Real-World Data
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Inha University Hospital (Other); Chonnam National University Hospital (Other); Nowon Eulji Medical Center (Unknown)
Responsible Party: Principal Investigator, Jung Hee Kim, Associate professor, Seoul National University Hospital
Other Study IDs: 2204-155-1320
Record Dates: First submitted 2024-01-05; First posted 2024-01-29 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Adrenal Tumor; Primary Aldosteronism; Cushing Syndrome; Pheochromocytoma; Adrenal Cortical Carcinoma
MeSH Terms: conditions — Adrenal Gland Neoplasms; Hyperaldosteronism; Cushing Syndrome; Pheochromocytoma; Adrenocortical Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Serum/Buffy coat to discover prognostic biomarkers and genetic background
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Nonfunctioning adrenal adenoma: Incidentally detected adrenal mass without hormone production
- Mild autonomous cortisol secretion: Adrenal tumors that do not meet the criteria for adrenal Cushing's syndrome but are not suppressed to below 1.8 µg/dL after the dexamethasone suppression test
- Adrenal Cushing syndrome: Adrenal diseases characterized by biochemical hypercortisolism accompanying with overt Cushingoid features.
- Primary aldosteronism: Adrenal diseases characterized by the excessive production of the hormone aldosterone and suppressed renin.
  Diagnostic criteria are as the following:
  1. Plasma aldosterone level of ≥6 ng/dL after a seated saline infusion test
  2. Plasma aldosterone level of ≥13 ng/dL after a captopril challenge test.
- Pheochromocytoma and paraganglioma: Chromaffin-originated tumors in the adrenal gland and others, characterized by catecholamine excess
- Adrenal cortical carcinoma: Malignant tumors originated from the adrenal cortex, which was confirmed by biopsy or pathology results

SUMMARY:
This research aims to establish clinical evidence for optimal treatment guidelines for adrenal diseases using real-world data. The approach involves building prospective and retrospective patient registries, which will be utilized to develop and conduct research on disease-specific protocols for adrenal disorders. The study targets patients with primary aldosteronism, pheochromocytoma, adrenal cancer, adrenal incidentalomas, and mild autonomous cortisol secretion. Registries for patients with adrenal diseases will be obtained from Seoul National University Hospital and Asan Medical Center, along with securing a common data model. The ultimate goal is to conduct research to generate clinical evidence for adrenal diseases using these resources.

DETAILED DESCRIPTION:
The ultimate goal is to develop clinical evidence for unmet needs in adrenal gland diseases using real-world data, thereby contributing to the optimization of treatment guidelines. This involves:

1. Generating real-world healthcare data through prospective and retrospective registries specific to each adrenal disease.
2. Acquiring a common data model for adrenal diseases, applicable across both domestic and international multicenter settings.
3. Creating real-world data linked with hospital medical records and public data for each adrenal disease, utilizing anonymized information merging services.
4. Developing and conducting research based on prospective and retrospective registries, a common data model, and the utilization of public-medical data for different adrenal diseases.

Study Design:

Prospective and retrospective patient registries.

Study Population:

Patients with adrenal gland disorders, including primary aldosteronism, pheochromocytoma, adrenal cancer, adrenal incidentalomas, and mild autonomous cortisol secretion

Research Methods:

1. Securing prospective and retrospective registries of patients with adrenal diseases.
2. Obtaining a common data model for adrenal diseases.
3. Utilizing the secured registries and common data model for multicenter studies to generate clinical evidence for adrenal diseases.
4. Linking public and medical data with the secured registries to further research in generating clinical evidence for adrenal diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients with adrenal diseases such as adrenal cortical carcinoma, Cushing's syndrome, primary aldosteronism, pheochromocytoma, adrenal incidentaloma
* patients who are 19 years or older

Exclusion Criteria:

* patients younger than 19 years old

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with adrenal disorders
Sampling Method: Non-Probability Sample
Enrollment: 8200 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of cardiovascular event | up to 20years
  Cardiovascular event

SECONDARY OUTCOMES:
Mortality rate | up to 20years
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hee Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided